CLINICAL TRIAL: NCT01286480
Title: Evaluation of Novel Transition Interventions for Youth With Congenital Heart Disease
Brief Title: Congenital Heart Adolescents: Program of Transition Evaluation Research
Acronym: CHAPTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other); Stollery Children's Hospital Foundation (Other)
Responsible Party: Principal Investigator, Andrew Mackie, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AM-Chapter-01
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Congenital Heart Defects
Keywords: Health Care Transition; Adolescent
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic-based Educational Intervention (Experimental): This will involve a 60 minute interaction between the teen and an advanced practice nurse (APN) in the cardiology clinic. A MyHealth passport will be created covering the name of the teen's cardiac condition, previous cardiac interventions, and name and purpose of the teen's medications. Potential late cardiac complications and contact names and location of local adult CHD cardiologists will also be reviewed. Three scenarios regarding adolescent risk taking behaviors (written in the 3rd person) will be presented to the teen who will be asked what advice he/she would offer to the teen in each of those scenarios. The teen will be given a study email address and encouraged to contact the APN by email or text messaging with follow-up questions. If no contact is initiated after 1 week, the APN will email or text (based on preference) the youth, to discuss additional questions.
  Interventions: Behavioral: Clinic-based Educational Intervention
- Usual Care (No Intervention): Youth seen in the Cardiology clinic see a nurse only to measure weight, height, and blood pressure. They rely on their cardiologist for information about their heart condition. The approach and amount of time taken by each cardiologist with a youth varies. Time-pressured clinic visits limit the opportunity to discuss many of the topics noted above.

INTERVENTIONS:
Behavioral: Clinic-based Educational Intervention — This will involve a 60 minute interaction between the teen and an advanced practice nurse (APN) in the cardiology clinic. A MyHealth passport will be created covering the name of the teen's cardiac condition, previous cardiac interventions, and name and purpose of the teen's medications. Potential late cardiac complications and contact names and location of local adult CHD cardiologists will also be reviewed. Three scenarios regarding adolescent risk taking behaviors (written in the 3rd person) will be presented to the teen who will be asked what advice he/she would offer to the teen in each of those scenarios. The teen will be given a study email address and encouraged to contact the APN by email or text messaging with follow-up questions. If no contact is initiated after 1 week, the APN will email or text (based on preference) the youth, to discuss additional questions.
  Arms: Clinic-based Educational Intervention

SUMMARY:
The objective of this study is to evaluate the potential role of a cardiology clinic-based educational intervention for 15 to 17 year olds with congenital heart disease (CHD) and their parents, and to determine whether this intervention results in improved self-management skills (e.g., renewing medication prescriptions), teens having greater knowledge of their heart condition, and more teen and parent satisfaction with services. The results of this study will form the basis for a website that in turn may serve as an additional means of providing transition interventions. The results of this study may also be applicable to youth with other special health care needs.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-17
* Followed in the Stollery Pediatric Cardiology Clinic or the Northern Alberta Adult Congenital (NAACH) clinic
* Moderate or Complex Congenital Heart Disease (as defined by the 2001 Bethesda guidelines) or Acquired Heart Disease (cardiomyopathy (dilated, hypertrophic, or restrictive forms), Marfan's syndrome or rheumatic heart disease with cardiac involvement)

Exclusion Criteria:

* Developmental Delay, reading level below grade 6 based on patient or parent report

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Mackie, MD, SM, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawicki GS, Lukens-Bull K, Yin X, Demars N, Huang IC, Livingood W, Reiss J, Wood D. Measuring the transition readiness of youth with special healthcare needs: validation of the TRAQ--Transition Readiness Assessment Questionnaire. J Pediatr Psychol. 2011 Mar;36(2):160-71. doi: 10.1093/jpepsy/jsp128. Epub 2009 Dec 29. PMID 20040605
- [Background] Warnes CA, Liberthson R, Danielson GK, Dore A, Harris L, Hoffman JI, Somerville J, Williams RG, Webb GD. Task force 1: the changing profile of congenital heart disease in adult life. J Am Coll Cardiol. 2001 Apr;37(5):1170-5. doi: 10.1016/s0735-1097(01)01272-4. No abstract available. PMID 11300418
- [Result] Mackie AS, Islam S, Magill-Evans J, Rankin KN, Robert C, Schuh M, Nicholas D, Vonder Muhll I, McCrindle BW, Yasui Y, Rempel GR. Healthcare transition for youth with heart disease: a clinical trial. Heart. 2014 Jul;100(14):1113-8. doi: 10.1136/heartjnl-2014-305748. Epub 2014 May 19. PMID 24842870

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: The intervention was conducted by one of three experienced cardiology nurses following intervention-facilitation training and fidelity assurance. The intervention involved a meeting with the nurse and the participant, with the exception of three interventions also attended by a father (n=1), an uncle (n=1) and a participant's friend (n=1). Interventions were held in a quiet room without other distractions, a short walk from the cardiology clinic. The order of the intervention was consistently followed, and the study nurse completed a log and field notes to document any difficulties that were encountered during the intervention and the participant's reaction, level of engagement, questions and body language. Interventions were offered on the same day as a routine clinic visit, or at a later date, depending on the participant's preference.
- Usual Care: Participants allocated to the usual care group were unaware of the intervention being offered to the treatment group. This was intended to prevent contamination by self-education or other means.
Period: Overall Study
Arm/Group | Intervention Arm | Usual Care
Started | 32 | 34
Completed | 27 | 31
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Population: We enrolled 66 participants. 5 intervention participants and 3 usual care participants withdrew their participation from the study before any study measures were completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinic-based Educational Intervention | Usual Care | Total
Number analyzed (Participants) | 27 | 31 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (1.0) | 16.4 (1.0) | 16.5 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 28
  Male | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Transition Readiness Assessment Questionnaire (TRAQ) Score
Description: The TRAQ is the most rigorously evaluated transition readiness questionnaire available and was developed in the USA. It has 29 items with two domains, self-management (16 items) and self-advocacy (13 ). The TRAQ is at a grade 5.7 reading level and uses a Likert scale. Each item is scored 1-5, with 1 being assigned for responses of "No, I do not know how" and a score of 5 assigned for responses of "Yes, I always do this when I need to." The TRAQ scores produced include an overall score and a subscale score. The overall score and the subscale scores are calculated simply by taking the average score across the items in the questionnaire (or subscale). The higher the score, the greater the perceived self-management or self-advocacy skills of the participant. The lower scores indicate the participant has a lower perceived level of self-management or self-advocacy.
Time Frame: Baseline, 1 month and 6 months
Population: The intervention involve a 60 minute interaction between the teen and an advanced practice nurse (APN) in the cardiology clinic. The youth in the usual care arm see a nurse for vitals. They rely on their cardiologist for information about their heart condition. The approach and amount of time taken by each cardiologist with a youth varies.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: This involves a 60 minute interaction between the teen and an advanced practice nurse (APN) in the cardiology clinic. A MyHealth passport is created covering the name of the teen's cardiac condition, previous cardiac interventions, and name and purpose of the teen's medications. Potential late cardiac complications and contact names and location of local adult CHD cardiologists are also reviewed. Three scenarios regarding adolescent risk taking behaviors (written in the 3rd person) are presented to the teen who will be asked what advice he/she would offer to the teen in each of those scenarios. The teen will be given a study email address and encouraged to contact the APN by email or text messaging with follow-up questions. If no contact is initiated after 1 week, the APN will email or text (based on preference) the youth, to discuss additional questions.
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 27 | 31
units on a scale
  Baseline Self-management | 2.77 (1.07) | 2.95 (0.98)
  Baseline Self-advocacy | 3.80 (0.79) | 3.92 (0.67)
  1 Month Self-management | 3.12 (0.75) | 3.08 (0.93)
  1 Month Self-advocacy | 4.03 (0.52) | 3.88 (0.75)
  6 Month Self-management | 3.59 (0.83) | 3.16 (1.05)
  6 Month Self-advocacy | 4.38 (0.56) | 4.01 (0.95)

2. Secondary Outcome: MyHeart Score
Description: Change in patient knowledge of his/her CHD (MyHeart score), comparing baseline to 1 month and 6 months follow-up. The MyHeart scale was developed for this study and has a grade 4.6 reading level. It consists of seven short answer or multiple-choice questions. Given the heterogeneity of prior medical and surgical interventions and need for medications in adolescents with heart disease, the denominator for some questions varied from one participant to the next. Accordingly, each participant was assigned a percentage correct score (numerator/denominator×100) at each time point. Higher percentage correct score reflects better patient knowledge of his/her CHD
Time Frame: Baseline, 1 month and 6 months
Measure: Mean (Standard Deviation); unit: percentage of score
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 27 | 31
percentage of score
  Baseline MyHeart score (%) | 57 (20) | 58 (25)
  1 Month MyHeart score (%) | 74 (15) | 61 (25)
  6 Month MyHeart score (%) | 75 (15) | 61 (25)

ADVERSE EVENTS:
Groups:
- Intervention: This will involve a 60 minute interaction between the teen and an advanced practice nurse (APN) in the cardiology clinic. A MyHealth passport will be created covering the name of the teen's cardiac condition, previous cardiac interventions, and name and purpose of the teen's medications. Potential late cardiac complications and contact names and location of local adult CHD cardiologists will also be reviewed. Three scenarios regarding adolescent risk taking behaviors (written in the 3rd person) will be presented to the teen who will be asked what advice he/she would offer to the teen in each of those scenarios. The teen will be given a study email address and encouraged to contact the APN by email or text messaging with follow-up questions. If no contact is initiated after 1 week, the APN will email or text (based on preference) the youth, to discuss additional questions.
- Usual Care: The youth in the usual care arm see a nurse for vitals. They rely on their cardiologist for information about their heart condition. The approach and amount of time taken by each cardiologist with a youth varies.
Arm/Group | Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/31
Other Adverse Events (participants affected / at risk) | 0/27 | 0/31

LIMITATIONS AND CAVEATS:
1. single centre trial
2. most interventions were conducted by a single nurse
3. assessed self-management behaviours based on self-report
4. long-term follow-up and attendance in an adult cardiac clinic were not assessed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes